CLINICAL TRIAL: NCT05114447
Title: RIsk Factors, Diagnosis, and Management of SEvere/Uncontrolled Asthma From General Population to Clinical Setting: Update and Follow-up of the RItA Registry
Brief Title: Severe/Uncontrolled Asthma From General Population to Clinical Setting: Update and Follow-up of the RItA Registry
Acronym: RISER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Pisa (Other)
Collaborators: University Hospital of Pisa (Unknown); National Research Council, Institute of Clinical Physiology, Italy (Other); University Of Perugia (Other); University Hospital of Ancona (Unknown)
Responsible Party: Principal Investigator, Laura Carrozzi, Full Professor of Medicine, University of Pisa
Other Study IDs: 213698
Record Dates: First submitted 2021-07-07; First posted 2021-11-10 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Asthma; Asthma Severe Persistent Uncontrolled
Keywords: risk factors; severe/uncontrolled asthma; clinical setting; general population; longitudinal study
MeSH Terms: conditions — Asthma | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical sample: a) clinical cases of severe/uncontrolled asthma attending hospital specialist centres already included in the online RItA Registry and b) new clinical cases of severe/uncontrolled asthma attending the clinical centres and not yet included in the online RItA Registry, with the following characteristics: adult subjects with a diagnosis of asthma since at least one year with a) uncontrolled asthma, despite regular treatment with GINA (Global Initiative for Asthma) step 4 level, in the last three months or b) controlled asthma with a step 5 level treatment according to GINA (Global Initiative for Asthma).
  Interventions: Other: Routine medical care
- Epidemiological sample: a) epidemiological cases of severe/uncontrolled asthma from a general population Pisa cohort already inserted in the online RItA Registry and b) new epidemiological cases of severe/uncontrolled asthma from pre-existing Pisa cohort not yet included in the online RItA Registry, with the following characteristics: adult subjects with at least one asthma attack in the last 12 months or wheezing and/or asthma therapy in the last 12months.
  Interventions: Other: Routine medical care; Other: Telephone interview

INTERVENTIONS:
Other: Routine medical care — Eligible subjects will be contacted from physicians, by telephone or directly when they attend the clinical centre for control visits. Once the patients have provided their signed informed consent, they will have to fill in the clinical form and to perform routine functional/clinical tests.
  Subjects will be investigated at baseline (T0), at 6-month follow-up (T6) and at 12-month follow-up (T12).
  All the possible variations that could occur in the patients' disease status and disease management, according to the routine medical care, will be registered and taken into account in the RISER study.
  RISER study is not a clinical trial, but it is an observational study without any specific drug administration by the investigators. Participants will receive interventions, which can include medical products, such as drugs or devices, or procedures, as part of their routine medical care but they will not be assigned to specific interventions by the investigator as in a clinical trial.
Other: Telephone interview — Eligible subjects will be contacted by telephone from trained personnel of the Research Unit. Once the signed informed consent is obtained by each enrolled subject, they will be invited to answer the phone questionnaire.
  Subjects will be investigated at baseline (T0) and at 12-month follow-up (T12). Subjects fitting the epidemiological definition of severe/uncontrolled asthma will be invited at the Pisa clinical centre to have routine clinical/functional tests.
  Each subject performing baseline clinical/functional tests at the Pisa clinical centre will be clinically and functionally re-assessed
  Groups: Epidemiological sample

SUMMARY:
Within the AGAVE project (2010-2014), funded by the 2008 AIFA (Italian Medicines Agency) Call (contract No. FARM8YRYZC), a severe/uncontrolled asthma online Registry (RItA) was implemented to assess the appropriateness of therapeutic strategies for severe/uncontrolled asthma patients, according to GINA (Global Initiative for Asthma) guidelines, in epidemiological and clinical samples. The online RItA Registry is a database containing information on patients' general characteristics, medical history, clinical data, risk factors, comorbidity, asthma exacerbations, current asthma treatment. Currently, it contains information on severe/uncontrolled asthma subjects, enrolled at national level, performing baseline (n tot=1018) and follow-up interviews (n tot=402).

Aim of the RISER study is to increase knowledge about the risk factors, diagnosis, and management of severe/uncontrolled asthma in general population and clinical setting through the update and follow-up of the RItA registry.

The RISER study is an observational longitudinal study involving a clinical setting and an epidemiological one.

The field survey will comprise one or two follow-ups according to the sample.

1. Observational longitudinal study in hospital specialist centres (clinical sample). Clinical cases of severe/uncontrolled asthma already included in the online RItA Registry and new clinical cases of severe/uncontrolled asthma attending the clinical centres and not yet included in the online RItA Registry, will be investigated at T0, T6 and T12 through a clinical form in order to collect information in accordance with the online RItA registry, and routine clinical/functional tests of asthma control.
2. Observational longitudinal study in a general population sample (epidemiological sample). Epidemiological cases of severe/uncontrolled asthma from Pisa cohort already inserted in the online RItA Registry and new epidemiological cases of severe/uncontrolled asthma from pre-existing Pisa cohort not yet included in the online RItA Registry will be investigated at T0 and T12 through a questionnaire to collect information for feeding the online RItA registry. Subjects fitting the epidemiological definition of severe/uncontrolled asthma will be invited at the Pisa clinical centre to have routine clinical/functional tests.

All data collected from clinical/epidemiological centres will be included in the RItA registry.

Overall, it is expected to enroll 422 patients.

DETAILED DESCRIPTION:
RISER study is an observational longitudinal study in epidemiological and clinical samples investigated through questionnaires/clinical forms and routine clinical/functional assessments at baseline and at follow-ups.

The study is constituted by two arms:

1. observational longitudinal study in hospital specialist centres (clinical sample);
2. observational longitudinal study in a general population sample (epidemiological sample).

The clinical sample will provide a new characterization of severe/uncontrolled asthma phenotypes through clinical and functional assessments and biomarkers.

The epidemiological sample will allow to obtain new information about risk/protective factors for severe/uncontrolled asthma and to identify new cases who have not been yet referred to clinical centres.

RISER study is not a clinical trial, but it is an observational study without any specific drug administration by the investigators. Participants will receive interventions, which can include medical products, such as drugs or devices, or procedures, as part of their routine medical care, but they will not be assigned to specific interventions by the investigator as in a clinical trial.

Sample size Considering a possible loss to follow-up and a refusal rate of 20%, the expected number of subjects in the clinical sample will be 287 (195 cases already included in the online RItA Registry and 92 new uncontrolled/severe asthma cases not yet included in the Registry).

Considering a possible loss to follow-up and a refusal rate of 30%, the expected number of subjects in the epidemiological sample will be 135 (112 cases already included in the online RItA Registry and 23 new uncontrolled/severe asthma cases not yet included in the Registry).

Data collection tools:

1. Clinical form (clinical sample): a modified and updated version of the RItA Registry implemented during the AGAVE study will be used;
2. Questionnaire (epidemiological sample): a modified and updated version of the questionnaire implemented during the AGAVE study will be used. The questionnaire will be structured according to the data required by the online RItA registry.

   The clinical form and the questionnaire will take into account the following aspects, as in the pre-existing RItA Registry: demographic characteristics, asthma severity and level of control, current asthma therapy, comorbidities, risk factors, health services utilization.

   New information, to answer to new specific aspects addressed in the RISER study, will be integrated: asthma indirect costs, quality of life, biological drugs use, reason of changing therapy, use of electronic cigarettes or of heat-not-burn tobacco.
3. Routine clinical /functional tests of asthma control (clinical and epidemiological sample):

serum total IgE, spirometry, reversibility test, blood cell count, fractional exhaled nitric oxide (FeNO), oscillometry.

Data collected from clinical and epidemiological centres will be included in the online RiTA registry.

Field survey The field survey will be organized in three or two phases, according to the type of sample. In particular, the field study will comprise T0, baseline, T6, follow-up at 6 months from baseline (only for the clinical sample), T12, follow-up at 12 months from baseline.

1. Observational longitudinal study in hospital specialist centres (clinical sample): eligible subjects will be contacted from physicians, by telephone or directly when they attend the clinical centre for control visits. Once the patients have provided their signed informed consent, they will have to fill in the clinical form; routine functional/clinical tests will be performed. In particular, subjects will be investigated at T0, T6 and T12 through the clinical form in order to collect information in accordance with the online RItA Registry and routine clinical/functional tests of asthma control.

   All the possible variations that could occur in the patients' disease status and disease management, according to the routine medical care, will be registered and taken into account in the RISER study.
2. Observational longitudinal study in a general population sample (epidemiological sample): eligible subjects will be contacted by telephone from trained personnel of the Research Unit.

Once the signed informed consent is obtained by each enrolled subject, they will be invited to answer the phone questionnaire and to perform a medical examination at the local clinical centre.

In particular, subjects will be investigated at T0 and T12 through the questionnaire to collect information for feeding the online RItA Registry. Subjects fitting the epidemiological definition of severe/uncontrolled asthma will be invited at the Pisa clinical centre (CC) to have routine clinical/functional tests.

Each subject performing baseline clinical/functional tests at the Pisa clinical centre (CC) will be clinically and functionally re-assessed.

. Statistical analysis: data quality control will be carried out before statistical analysis performance.

Descriptive analysis will comprise: frequency distribution and Chi-square test for categorical variables; analysis of variance and Wilcoxon's rank test for continuous variables.

Multivariable analysis will be carried out through logistic regression analysis and survival analysis, taking into account the independent effects of potential confounders. Analyses to assess asthma phenotypes/endotypes and presence of risk factors clusters will be performed (i.e. cluster analysis, network analysis, principal component analysis) as well.

Analysis on cross-sectional and longitudinal data will be carried out. The longitudinal analysis will take into account a follow-up period of 6 and 12 months. For subjects already included in the online RItA Registry, a longer follow-up will be assessed (from 5 to 9 years).

Comparisons between the different phases of the study will permit to collect information about changes in asthma condition; in particular, the following statistical analysis will be carried out:

1. assessment of incidence and prevalence of severe/uncontrolled asthma and related risk factors in asthmatic cohorts;
2. comparison between different therapeutic approaches and related effectiveness in terms of asthma control, in the whole sample and taking into account comorbidity and polypharmacy;
3. assessment of possible risk factors for severe/uncontrolled asthma (i.e. demographic characteristics, environmental/occupational exposure, comorbidity) related to a different effectiveness of the therapeutic approach;
4. assessment of treatable traits related to different effectiveness of the therapeutic approach;
5. assessment of severe/uncontrolled asthma average indirect costs, in the whole sample and in specific subgroups of patients, in relation to gender, age, environmental exposures, comorbidity;
6. assessment of risk factors (i.e. demographic characteristics, environmental/occupational exposure, comorbidity) related to different disease prognosis;
7. characterization of specialist clinical setting and epidemiological setting in terms of risk factors exposure, therapeutic approaches and asthma control;
8. assessment of characteristics of new cases, enrolled from the epidemiological cohort and clinically confirmed, who have not been yet referred to clinical centres.

Ethical aspects: No issue about the safety of the protocol has to be forecasted, since all the protocol procedures are routine analyses for severe/uncontrolled asthma patients.

Study subjects will not undergo any risk for their physical or psychological domains, as they will perform questionnaire interview and a regular medical examination under safe procedures.

According to the General Data Protection Regulation (GDPR 25 May 2018), informed consent for data collection and analysis will be requested to the subjects involved in the study.

ELIGIBILITY:
Inclusion Criteria

1. Observational longitudinal study in hospital specialist centres (clinical sample) Target population consists of asthmatic adult patients managed by clinical centres in Pisa (Unit of Pulmonology, Cardio-Thoracic and Vascular Department), Perugia (Section of Occupational Medicine, Respiratory Diseases and Toxicology, Medicine Department), Ancona (Unit of Allergology, Internal Medicine Department).

   In particular, the eligible patients for RISER study are:
   1. clinical cases of severe/uncontrolled asthma already included in the online RItA Registry (number: 244 total; n=75 Pisa; n=114 Perugia; n=55 Ancona)
   2. new clinical cases of severe/uncontrolled asthma attending the clinical centres and not yet included in the online RItA Registry, with the following characteristics: adult subjects with a diagnosis of asthma since at least one year with a) uncontrolled asthma, despite regular treatment with GINA step 4 level, in the last three months or b) controlled asthma with a step 5 level treatment according to GINA. The expected number will be of 115 in total: n=50 Pisa; n=35 Perugia; n=30 Ancona.
2. Observational longitudinal study in a general population sample (epidemiological sample) Target population consists of adults suffering from asthmatic symptoms or having an asthma diagnosis within a general population sample investigated in three subsequent cross-sectional surveys in Pisa (the 1st survey (PI1) performed in 1985-1988 on 3865 subjects; the 2nd survey(PI2) in 1991-1993 on 2841 subjects; the 3rd survey (PI3) in 2009-2011 on 1620 subjects).

In particular, the eligible subjects for RISER study are:

1. epidemiological cases of severe/uncontrolled asthma from Pisa cohort already inserted in the online RItA Registry (n=160)
2. new epidemiological cases of severe/uncontrolled asthma from pre-existing Pisa cohort not yet included in the online RItA Registry, with the following characteristics: adult subjects with at least one asthma attack in the last 12 months or wheezing and/or asthma therapy in the last 12 months. The expected number, on the basis of the severe/uncontrolled asthma prevalence obtained in previous studies, is 34.

Exclusion Criteria

1. subjects of age < 18 yrs
2. subjects unable to participate in the study or to sign the consent form
3. subjects refusing to fill in the consent form
4. untraceable subjects (for the epidemiological sample)

No other specific exclusion criterion will be considered, in order to capture all potential variables influencing severe/uncontrolled asthma outcomes in real life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Severe/uncontrolled asthma patients managed by clinical centres in Pisa (Unit of Pulmonology, Cardio-Thoracic and Vascular Department), Perugia (Section of Occupational Medicine, Respiratory Diseases and Toxicology, Medicine Department), Ancona (Unit of Allergology, Internal Medicine Department).
  2. Severe/uncontrolled asthma subjects from a pre-existing cohort of general population living in Pisa.
Sampling Method: Non-Probability Sample
Enrollment: 422 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change of asthma control test (score) | Analyzed at baseline, month 6 and month 12.
  - asthma control test - ACT (score range 5-25, with higher scores indicating greater asthma control) (mean score)
Change of asthma control questionnaire (score) | Analyzed at baseline, month 6 and month 12.
  - asthma control questionnaire - ACQ (score range 0- 6, with lower scores indicating greater asthma control) (mean score)
Change of asthma exacerbations (number) | Analyzed at baseline, month 6 and month 12.
  - asthma exacerbations (mean number)
Change of use of systemic steroids (number) | Analyzed at baseline, month 6 and month 12.
  - systemic steroids (number of courses)
Change of use of biologic therapy (number) | Analyzed at baseline, month 6 and month 12.
  - biologic therapy (number of months)

SECONDARY OUTCOMES:
Health services use-hospitalization | Analyzed at baseline, month 6 and month 12.
  - hospitalization (number of hospitalization due to asthma)
Health services use-emergency department visits | Analyzed at baseline, month 6 and month 12.
  - emergency department (ED) visit (number of ED visits due to asthma)
Impairment of work/school (number) | Analyzed at baseline, month 6 and month 12.
  - work/school absenteeism (number of days)
Impairment of other daily activities (number) | Analyzed at baseline, month 6 and month 12.
  - limitations in daily activities (number of days)
Quality of life (score) | Analyzed at baseline, month 6 and month 12.
  Quality of life score (Asthma Quality of Life Questionnaire; global score range 1-7 with higher scores indicating better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Carrozzi, MD, Principal Investigator — University of Pisa
Locations (4):
- Italy (4):
  - Leonardo Antonicelli, Ancona
  - Nicola Murgia, Perugia
  - Laura Carrozzi, Pisa
  - Sandra Baldacci, Pisa

IPD SHARING:
Plan to Share IPD: No
Only researchers involved in the RISER study will have access to the individual participant data.

REFERENCES:
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Pavord ID, Beasley R, Agusti A, Anderson GP, Bel E, Brusselle G, Cullinan P, Custovic A, Ducharme FM, Fahy JV, Frey U, Gibson P, Heaney LG, Holt PG, Humbert M, Lloyd CM, Marks G, Martinez FD, Sly PD, von Mutius E, Wenzel S, Zar HJ, Bush A. After asthma: redefining airways diseases. Lancet. 2018 Jan 27;391(10118):350-400. doi: 10.1016/S0140-6736(17)30879-6. Epub 2017 Sep 11. No abstract available. PMID 28911920
- [Background] McDonald VM, Hiles SA, Godbout K, Harvey ES, Marks GB, Hew M, Peters M, Bardin PG, Reynolds PN, Upham JW, Baraket M, Bhikoo Z, Bowden J, Brockway B, Chung LP, Cochrane B, Foxley G, Garrett J, Jayaram L, Jenkins C, Katelaris C, Katsoulotos G, Koh MS, Kritikos V, Lambert M, Langton D, Lara Rivero A, Middleton PG, Nanguzgambo A, Radhakrishna N, Reddel H, Rimmer J, Southcott AM, Sutherland M, Thien F, Wark PAB, Yang IA, Yap E, Gibson PG. Treatable traits can be identified in a severe asthma registry and predict future exacerbations. Respirology. 2019 Jan;24(1):37-47. doi: 10.1111/resp.13389. Epub 2018 Sep 19. PMID 30230137
- [Background] Peters SP, Ferguson G, Deniz Y, Reisner C. Uncontrolled asthma: a review of the prevalence, disease burden and options for treatment. Respir Med. 2006 Jul;100(7):1139-51. doi: 10.1016/j.rmed.2006.03.031. Epub 2006 May 18. PMID 16713224
- [Background] Novelli F, Latorre M, Vergura L, Caiaffa MF, Camiciottoli G, Guarnieri G, Matucci A, Macchia L, Vianello A, Vultaggio A, Celi A, Cazzola M, Paggiaro P; Xolair Italian Study Group. Asthma control in severe asthmatics under treatment with omalizumab: a cross-sectional observational study in Italy. Pulm Pharmacol Ther. 2015 Apr;31:123-9. doi: 10.1016/j.pupt.2014.09.007. Epub 2014 Sep 30. PMID 25281265
- [Background] Farne HA, Wilson A, Powell C, Bax L, Milan SJ. Anti-IL5 therapies for asthma. Cochrane Database Syst Rev. 2017 Sep 21;9(9):CD010834. doi: 10.1002/14651858.CD010834.pub3. PMID 28933516
- [Background] Varsano S, Segev D, Shitrit D. Severe and non-severe asthma in the community: A large electronic database analysis. Respir Med. 2017 Feb;123:131-139. doi: 10.1016/j.rmed.2016.12.017. Epub 2016 Dec 28. PMID 28137489
- [Background] Maio S, Baldacci S, Bresciani M, Simoni M, Latorre M, Murgia N, Spinozzi F, Braschi M, Antonicelli L, Brunetto B, Iacovacci P, Roazzi P, Pini C, Pata M, La Grasta L, Paggiaro P, Viegi G; AGAVE group. RItA: The Italian severe/uncontrolled asthma registry. Allergy. 2018 Mar;73(3):683-695. doi: 10.1111/all.13342. Epub 2017 Nov 22. PMID 29072882
- [Background] Adachi M, Kozawa M, Yoshisue H, Lee Milligan K, Nagasaki M, Sasajima T, Miyamoto T, Ohta K. Real-world safety and efficacy of omalizumab in patients with severe allergic asthma: A long-term post-marketing study in Japan. Respir Med. 2018 Aug;141:56-63. doi: 10.1016/j.rmed.2018.06.021. Epub 2018 Jun 28. PMID 30053973